CLINICAL TRIAL: NCT05202431
Title: The Effect of Telephone Follow-up and Training on Treatment Adherence in Tuberculosis Patients and Contacts: A Randomised, Controlled and Quasi Experimental Study
Brief Title: The Effect of Telephone Follow-up and Training on Treatment Adherence in Tuberculosis Patients and Contacts
Acronym: Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuberculosis Network European Trialsgroup (Network)
Responsible Party: Principal Investigator, Sema Aytaç, PhD, PhD, Tuberculosis Network European Trialsgroup
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TBNET
Record Dates: First submitted 2021-12-14; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Tuberculosis
Keywords: nursing education; tuberculosis; tuberculosis contact; treatment adherence; telephonefollow-up
MeSH Terms: conditions — Tuberculosis; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adherence (Experimental): Participants received training, telefollow-up and daily text messages for 6 months.
  Interventions: Behavioral: Treatment adherence
- Standart care (No Intervention): The standard follow-up applied in the dispensary for this group was performed.

INTERVENTIONS:
Behavioral: Treatment adherence — The patients were reminded to take drug by patient training, telephone follow-up, and daily sms. It was determined that the effect of the training and telephone follow-up provided to the TB patients and contacts on the treatment adherence.
  Arms: Adherence

SUMMARY:
Tuberculosis (TB) is a preventable and curable disease mostly affecting lungs and caused by the bacteria called as Mycobacterium Tuberculosis (MTB). It is estimated that approximately 10 million people are diagnosed with TB every year in the world and 1.7 billion people are infected by MTB and at risk in terms of the development of the disease. Contacted person is the one who shares the same environment with the patient suffering from contagious TB and is exposed to MTB bacilli.

Today, the aim of the TB control and prevention programs is to determine the active TB patients and provide cure by healing and also to screen those contacted with the TB patients and determine whether or not they have latent TB infection and treat them and to detect the active cases among the contacts. In the current guidelines, the importance of screening all the contacts of the patients with pulmonary TB and applying a protective treatment for the household in terms of community health care is emphasised. For this reason, it is of prime importance to perform contact screening of the relatives of the TB patients and apply protective treatment. The patients receiving TB and TB protection treatment need to use medicine regularly for at least six months. It is highly important to adherence this period for the success of the treatment. However, it has been reported in the literature that the rate of nonadherence to the TB treatment varies between 20-80% and the nonadherence to the TB treatment is the most serious barrier in the control of the disease. İncomplete treatment may result in long-lasting infection, drug resistance, relapse, and death.

In the litareture, it has been stated in the study conducted with the individuals with some chronic diseases that tele-follow-up is effective in providing the self-care agency of patients and the cognitive-social adaptation. It has been reported that some problems emerge especially in the TB patients such as the interruption of treatment, forgetting medication (24.5%), side-effects of drugs, (23.3%), symptomatic recovery (19.5%), failure to know the necessity of completing the life cycle of drugs by most of patients and not receiving adequate training and these problems may be managed more effectively by tele-follow-up.

As is known, nurses are involved in all the processes of protecting-promoting the health of the individuals, families and society and their recovery in case of disease. Moreover, providing the protective treatment by performing the required screening for treating TB patients, their follow-up and preventing the development of disease in contacted ones has a vital importance in preventing the spread of TB in the society. Nurses may follow the findings of patients, obtain information about the process, produce information and transmit information with this system (reporting drug changes, performing training follow-up of patients etc.). In the literature, it has been emphasised that tele-mobile nursing services is a cost-effective method since it decreases the hospitalisation rate and period of the TB patients. Accordingly, the main aim of this study is to assess the effect of the training and the telephone follow-up provided by the nurse for the TB patients and contacts on the medication adherence.

DETAILED DESCRIPTION:
This research was conducted as a randomised, controlled and quasi-experimental study to determine the effect of the training and telephone follow-up provided to the TB patients and contacts on the treatment adherence. The population of the study was composed of the patients receiving treatment in a tuberculosis control dispensary between July 2018-July 2019. The sample size was calculated to be 28 in each group through power analysis. Eighty-one TB patients and 90 TB contacts were included in the study. However, 15 TB patients and 3 contacts were excluded since they were transferred to another dispensary and they died. The study was completed with 66 TB patients in the intervention (n= 32) and control groups (n=34) and 87 contacts in the intervention (n= 41) and control groups (n = 46) The TB patients who applied to the dispensary and their contacts were informed about the aim and scope of the study. Then, four groups were formed by using the randomisation menu of the computer program: the intervention and control groups for the TB patients and the intervention and control groups for the contacts. The randomisation was conducted by a statistics specialist who had no contact with the participants. All participants were blinded to the randomisation procedure. However, the researchers were not blinded to the patient groups, due to the nature of the intervention.

The interviews were performed by using the face-to-face interview technique in the outpatient clinic. In the first interview, the questionnaire was applied to four groups; TB intervention and TB control group, Contact intervention and Contact control group.

ELIGIBILITY:
Inclusion Criteria:

* With pulmonary TB
* Being voluntary to participate in the study
* Being at and over the age of 18
* Having no communication problems
* Being able to use mobile telephone

Exclusion Criteria:

* Being under 18 years old
* Not voluntary to participate in the study
* Having multi drug resistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Change in treatment adherence during the Follow-up | 6 months
  Tuberculosis Adherence Determination Questionnaire (TADQ) was conducted. It is a 5-point likert scale and minimum and maximum scores of the scale are 26 and 175 and high score signifies that adherence increases.

CONTACTS AND LOCATIONS:
Overall Officials: Sema Aytac, Principal Investigator — Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aytac S, Ovayolu O, Dogru S. The effect of breathing exercises on fatigue in tuberculosis patients: a randomized controlled trial. Rev Assoc Med Bras (1992). 2024 Dec 2;70(12):e20240888. doi: 10.1590/1806-9282.20240888. eCollection 2024. PMID 39630726